CLINICAL TRIAL: NCT06905275
Title: A Phase 1 Clinical Trial to Evaluate the Safety and Immunogenicity of Glycan-trimmed HIV-1 Nanoparticle Vaccine (UVAX-1107), Followed by Homologous or Wild-type HIV-1 Nanoparticle Vaccine (UVAX-1197) Boost, Each Adjuvanted With 3M-052-AF + Alum in Adult Participants Without HIV
Brief Title: A Clinical Trial to Evaluate the Safety and Immunogenicity of Glycan-trimmed HIV-1 Nanoparticle Vaccine (UVAX-1107), Followed by Homologous or Wild-type HIV-1 Nanoparticle Vaccine (UVAX-1197) Boost, Each Adjuvanted With 3M-052-AF + Alum in Adult Participants Without HIV
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: Temporarily Closed (Paused) to Accrual
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 319; 39136 (Other: DAIDS DOCUMENT ID)
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-07

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — aluminum sulfate

STUDY DESIGN:
Intervention Model Description: The trial will begin with enrollment of Group 1. Groups 2 and 3 will open to enrollment concurrently. Enrollment in Group 2 and Group 3 will be randomized.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Treatment: 150 mcg of UVAX-1107 admixed with 5 mcg of 3M-052-AF + 500 mcg of Alum, to be administered at Weeks 0 and 8.
  Followed by: 150 mcg of UVAX-1197 admixed with of 5 mcg of 3M-052-AF + 500 mcg Alum to be administered at Weeks 20 and 32.
  Interventions: Biological: 3M-052-AF + Alum; Biological: UVAX-1107; Biological: UVAX-1197
- Group 2 (Experimental): Treatment: 300 mcg of UVAX-1107 admixed with 5 mcg of 3M-052-AF + 500 mcg of Alum to be administered at Weeks 0 and 8.
  Followed by: 300 mcg of UVAX-1197 admixed with 5 mcg of 3M-052-AF + 500 mcg of Alum to be administered at Weeks 20 and 32.
  Interventions: Biological: 3M-052-AF + Alum; Biological: UVAX-1107; Biological: UVAX-1197
- Group 3 (Experimental): Treatment: 300 mcg of UVAX-1107 admixed with 5 mcg of 3M-052-AF + 500 mcg of Alum to be at Weeks 0, 8, 20, and 32.
  Interventions: Biological: 3M-052-AF + Alum; Biological: UVAX-1107

INTERVENTIONS:
Biological: 3M-052-AF + Alum — Intramuscular (IM) injection
Biological: UVAX-1107 — IM injection
  Other Names: Glycan-trimmed
Biological: UVAX-1197 — IM injection
  Other Names: Wild Type (WT)
  Arms: Group 1; Group 2

SUMMARY:
This is a phase 1, first-in-human (FIH) trial for the combination of UVAX-1107 and UVAX-1197, both adjuvanted with 3M-052-AF + Aluminum Hydroxide Suspension (Alum). This means it is the first time this combination of study products is being tested in people.

The purpose of this study is to see if the study products are safe, if people are able to take them without becoming too uncomfortable, and how a person's immune system responds to them (a person's immune system protects them from infections and disease).

Twenty-five volunteers without HIV and in overall good health will be enrolled and be in this study for a little over 1 year (56 weeks) of clinic visits (about 12 visits), with a follow-up contact 1 year after the final injection to check on their health.

Study procedures will include blood draws, injections, and the collection of white blood cells and cells from their lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* Understand the study and agree to participate.
* Be available for follow-up visits and contact for 12 months after the last study product is administered.
* Be willing to undergo all study procedures.
* Not be in another study unless approved by both study sponsors.
* Be in good general health.
* Have normal physical exam and lab results.
* Agree to discuss HIV risk and prevention.
* Have a certain minimum hemoglobin level (≥ 11.0 g/dL for women, ≥ 13.0 g/dL for men).
* Have a white blood cell count within 2500 to 12,000/mm³.
* Have a platelet count between 125,000 to 550,000/mm³.
* Have an ALT level less than 2.5 times the upper limit of normal.
* Have a serum creatinine level within 1.1 times the normal limit.
* Have a serum calcium level of at least 8.5 mg/dL.
* Have blood pressure within specified limits.
* Test negative for HIV.
* Test negative for Hepatitis C.
* Test negative for Hepatitis B.
* Women who can become pregnant must use effective contraception and test negative for pregnancy at enrollment.
* Women who can become pregnant must agree not to seek pregnancy through alternative methods during the study period.

Exclusion Criteria:

* Breastfeeding or pregnant.
* BMI is 40 or higher (exceptions can be made if you're in good health).
* Diagnosed with diabetes (unless it's well-controlled Type 2 diabetes or gestational diabetes).
* Received an investigational HIV vaccine or monoclonal antibodies.
* Received a non-HIV investigational vaccine in the past year (exceptions exist for licensed or emergency-authorized vaccines).
* Have an immune deficiency or are taking medications that impair immune response.
* Received blood products or immunoglobulins within the last 16 weeks.
* Received certain vaccines within 4 weeks before enrollment.
* Received other vaccines within 14 days before enrollment.
* Started allergy immunotherapy within the last year (stable therapy is okay).
* Taken investigational research agents recently.
* Had a serious reaction to any vaccine.
* Have hereditary or acquired angioedema.
* Had unexplained hives in the past year.
* Have a bleeding disorder that would make study procedures risky.
* Had seizures or taken seizure medication in the past 3 years.
* Spleen has been removed or spleen doesn't work properly.
* Active duty or reserve US military personnel.
* Any serious health condition that could affect safety, rights, or ability to participate (including substance use, psychiatric disorders, recent suicide attempts, or cancer with potential recurrence).
* Asthma that requires frequent or high-dose medication, emergency care, or multiple maintenance therapies.
* History of certain immune-mediated medical conditions (mild, localized conditions may be okay).
* Allergic to local anesthetics like Novocaine or Lidocaine.
* History of difficult venous access or intravenous drug use.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-07-20 (Estimated); Study Completion 2027-07-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of local reactogenicity signs and symptoms | 56 weeks (collected for a minimum of 14 days following receipt of any study vaccine)
Incidence of systemic reactogenicity signs and symptoms | 56 weeks (collected for a minimum of 14 days following receipt of any study vaccine)
Number of participants experiencing Serious Adverse Events (SAEs) leading to early participant withdrawal or permanent discontinuation from the study | 108 weeks (throughout the study and for 52 weeks following any receipt of study product)
Number of participants experiencing Medically Attended Adverse Events (MAAEs) leading to early participant withdrawal or permanent discontinuation from the study | 108 weeks (throughout the study and for 52 weeks following any receipt of study product)
Number of participants experiencing Adverse Events of Special Interest (AESIs) leading to early participant withdrawal or permanent discontinuation from the study | 108 weeks (throughout the study and for 52 weeks following any receipt of study product)
Number of participants experiencing Adverse Events (AEs) leading to early participant withdrawal or permanent discontinuation from the study | 108 weeks (throughout the study and for 52 weeks following any receipt of study product)
Response rate of serum HIV-1 IgG binding antibodies against vaccine-matched Env antigens | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Assessed by binding antibody multiplex assay (BAMA)
Magnitude of serum HIV-1 IgG binding antibodies against vaccine-matched Env antigens | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Assessed by BAMA
Response rate of serum antibody (Ab) neutralization of tier 1 HIV-1 strains | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Measured by TZM-bl assay
Magnitude of serum Ab neutralization of tier 1 HIV-1 strains | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Measured by TZM-bl assay
Response rate of serum Ab neutralization of vaccine-matched tier 2 HIV-1 strains | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Measured by TZM-bl assay
Magnitude of serum Ab neutralization of vaccine-matched tier 2 HIV-1 strains | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Measured by TZM-bl assay

SECONDARY OUTCOMES:
Response rate of serum HIV-1 IgG binding antibodies against heterologous Env antigens | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Assessed by BAMA
Magnitude of serum HIV-1 IgG binding antibodies against heterologous Env antigens | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Assessed by BAMA
Magnitude-breadth of serum HIV-1 IgG binding antibodies against heterologous Env antigens | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Assessed by BAMA
Response rate of serum Ab neutralization of heterologous HIV-1 strains | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Measured by TZM-bl assay
Magnitude of serum Ab neutralization of heterologous HIV-1 strains | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Measured by TZM-bl assay
Response rate of epitope-specific binding | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Measured by electron microscopy polyclonal epitope mapping (EMPEM)
Response rate of Env-specific IgG+ B-cells | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Measured by flow cytometry analysis
Magnitude of Env-specific IgG+ B-cells | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Measured by flow cytometry analysis
Response rate of CD4+ T-cell responses | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Measured by intracellular cytokine staining
Magnitude of CD4+ T-cell responses | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Measured by intracellular cytokine staining
Response rate of CD8+ T-cell responses | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Measured by intracellular cytokine staining
Magnitude of CD8+ T-cell responses | Week 22 and Week 34 (2 weeks after the third and fourth vaccinations)
  Measured by intracellular cytokine staining
Response rate of serum HIV-1 IgG binding antibodies | Week 56 (24 weeks after the fourth vaccinations)
  Assessed by BAMA
Magnitude of serum HIV-1 IgG binding antibodies | Week 56 (24 weeks after the fourth vaccinations)
  Assessed by BAMA
Response rate of serum Ab neutralization | Week 56 (24 weeks after the fourth vaccinations)
  Measured by TZM-bl assay
Magnitude of serum Ab neutralization | Week 56 (24 weeks after the fourth vaccinations)
  Measured by TZM-bl assay
Response rate of Env-specific IgG+ B-cells | Week 56 (24 weeks after the fourth vaccinations)
  Measured by flow cytometry analysis
Magnitude of Env-specific IgG+ B-cells | Week 56 (24 weeks after the fourth vaccinations)
  Measured by flow cytometry analysis

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Alabama CRS (#31788), Birmingham, Alabama
  - Columbia P&S CRS (#30329), New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Vanderbilt Vaccine (VV) CRS (#30352), Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No